CLINICAL TRIAL: NCT06988709
Title: Examining the Most Effective Method to Reduce Running Ground Contact Time
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jennah Bulen, Principal Investigator, Keller Army Community Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KACH.2025.0009; 24KACH008 (Other: Keller)
Record Dates: First submitted 2025-04-18; First posted 2025-05-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Healthy Runners
Keywords: running; ground; gait; retraining; contact; time

STUDY DESIGN:
Intervention Model Description: Within-subjects, repeated measures design completed in a single session
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Run Retraining Conditions (Experimental): Single-arm, within subject, repeated measures design. All participants will run at baseline and then under 3 different running conditions.
  Interventions: Other: Real-time Visual Feedback; Other: Real-time Auditory Feedback; Other: Real-time Verbal Feedback

INTERVENTIONS:
Other: Real-time Visual Feedback — Runners will visualize their real-time ground contact time (GCT) measured by the RunScribe on a TV screen. They will be instructed to run with a goal of matching their target GCT. Their target GCT will be 5% less than their baseline.
Other: Real-time Auditory Feedback — Runners will be instructed to match their step rate to a target step rate, 10% above their baseline step rate. A metronome will be played over a speaker to provide real-time auditory feedback of the target step rate.
Other: Real-time Verbal Feedback — The clinician will provide real-time verbal feedback to runner to "pull your foot off the ground as quickly as you can," every 15 seconds during the retraining condition.

SUMMARY:
The purpose of our study is to establish the most effective running retraining technique to decrease ground contact time. This will be investigated by applying three running retraining conditions and assessing the change in ground contact time and other biomechanical variables between the runner's baseline running and each retraining technique.

DETAILED DESCRIPTION:
The purpose of our study is to establish the most effective running retraining technique to decrease ground contact time utilizing three common running retraining methods in healthy runners.

The first aim will be to apply three running retraining conditions and assess the change in ground contact time and other spatiotemporal and biomechanical variables between the runner's baseline running and each retraining condition.

The three running conditions will be at the participant's self-selected speed corresponding to "a comfortable run for 30 minutes". The conditions will be, condition 1: a verbal cue to "pull your foot off the ground as quickly as you can," condition 2: a metronome set to 10% above their preferred cadence found during the baseline run, and condition 3: visual feedback to reduce their ground contact time through observing that number in real time provided by a commercial IMU. The participant will attempt to lower that to 5% below their baseline run ground contact time by being given that target number on a sheet of paper.

The second aim will be to examine the effect of the 3 running conditions on the runner's level of exertion and difficulty using the Omni Rate of Perceived Exertional Scale, the Rate of Perceived Difficulty, and ranking the techniques from 1 to 3 on which they felt was most natural.

We hypothesize that each method will reduce ground contact time, but condition 3 providing continuous visual feedback will result in the most consistent decrease to ground contact time across the runners and will be perceived as the easiest to perform.

Overall, this study will provide clinicians with a running retraining intervention that has been objectively shown to decrease ground contact time and provide researchers with a method to further investigate its effect on running injuries.

ELIGIBILITY:
Inclusion Criteria:

* Military Service Member or USMA cadet between the ages of 17-60
* Run at least 2 miles three times per week for the past 3 months
* Able to run for at least 15 continuous minutes at a self-selected speed
* Fluent in the English language to read and provide informed consent and follow study instructions

Exclusion Criteria:

* Lower extremity or low back pain in the previous 3 months
* Lower extremity or low back surgery in the previous 6 months
* Self-reported pregnancy or given birth within the last 6 months
* Currently on a profile that restricts or limits running

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Ground Contact Time | Within a single session, measured pre-intervention (baseline) and during each running condition intervention
  The amount of time in milliseconds that the foot remains in contact with the ground while running. GCT will be measured through the RunScribe device.

SECONDARY OUTCOMES:
Step Rate | Within a single session, measured pre-intervention (baseline) and during each running condition intervention
  Number of steps per minute that the participant takes in one minute while running.
Average Vertical Loading Rate (AVLR) | Within a single session, measured pre-intervention (baseline) and during each running condition intervention
  Measured in Bodyweights/second. Total interval considered for loading rate is the start of stance phase through the impact peak location. We will calculate the average loading rate from 20% of the impact peak value to 80% of the impact peak magnitude.
Braking Impulse | Within a single session, measured pre-intervention (baseline) and during each running condition intervention
  Kg*m/s. The impulse associated with the deceleration while running.
Step Length | Within a single session, measured pre-intervention (baseline) and during each running condition intervention
  The distance measured in centimeters while running from one foot strike to the next foot strike.

CONTACTS AND LOCATIONS:
Locations (1):
- Keller Army Community Hospital, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: No
We do not have a data sharing agreement or plan to share IDP as part of our IRB protocol.